CLINICAL TRIAL: NCT04869969
Title: Supine Versus Prone Percutaneous Nephrolithotomy in the Pediatric Age Group? A Randomized Controlled Trial.
Brief Title: Supine Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R32/ 2019
Record Dates: First submitted 2021-03-06; First posted 2021-05-03 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Nephrolithotomy, Percutaneous; Supine Position; Prone Position

STUDY DESIGN:
Intervention Model Description: percutaneous nephrolithotomy to be performed in both supine and prone position
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and the statistician were blinded to the type of the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supine percutaneous nephrolithotomy (Experimental): percutaneous nephrolithotomy to be done in the supine position
  Interventions: Procedure: percutaneous nephrolithotomy (supine position)
- prone percutaneous nephrolithotomy (Active Comparator): percutaneous nephrolithotomy to be done in the prone position
  Interventions: Procedure: percutaneous nephrolithotomy ( prone position)

INTERVENTIONS:
Procedure: percutaneous nephrolithotomy (supine position) — percutaneous nephrolithotomy to be done in the supine position
  Arms: supine percutaneous nephrolithotomy
Procedure: percutaneous nephrolithotomy ( prone position) — percutaneous nephrolithotomy in the prone position
  Arms: prone percutaneous nephrolithotomy

SUMMARY:
there is an increased incidence of renal stones, especially in the pediatric age group. the percutaneous approach in the pediatric age took a long time till it again accepted among surgeons worldwide. the prone position is the preferred approach to perform percutaneous nephrolithotomy in the pediatric age group. this study aims to compare supine versus prone position percutaneous nephrolithotomy in the pediatric age group.

DETAILED DESCRIPTION:
The incidence of renal stones in the pediatric age group increased from 18.4 to 57.0% per100,000 children in the period from 1999 to 2008. The acceptance of PCNL in pediatrics was slow at first due to concerns of the small kidney size compared to relatively large instruments percutaneous nephrolithotomy in pediatric patients was conventionally performed in the prone position for historical reasons, being more familiar to surgeons and it was considered safer to avoid colonic injury.

Supine PCNL has several valuable advantages to pediatric patients in particular better irrigation shorter operative time with a comparable outcome with the prone position.

our study aims to assess the efficacy and the safety of percutaneous nephrolithotomy in the supine position in comparison to the prone position in the pediatric age group.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from two to sixteen years old with single or multiple renal stones indicated for percutaneous nephrolithotomy

Exclusion Criteria:

* patients with renal anomalies, bleeding tendency, elevated kidney function tests for age, previous renal surgical intervention on the same site of intervention.
* patients with skeletal abnormalities and spine deformities were also excluded
* patients with a single kidney were also excluded

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
stone free rate | first day postoperative
  evaluation of our patients after surgery with Xray or CT to detect residual stones

SECONDARY OUTCOMES:
Fluoroscopy time during the procedure in minutes | intraoperative finding in minutes,
  time of fluoroscopy exposure in minutes intraoperative, time of radiational exposure during the surgery. operative finding only
operative time of the procedure in minutes | intraoperative finding in minutes,
  time from patient positioning till the end of the procedure, operative finding only
rate of Hemoglobin drop | day 1 post operative
  change in the perioperative hemoglobin level
hospital stay | first 2 days post surgery
  days of hospital stay after the surgery
incidence of urinary tract infection | first 7 days post surgery
  presence of manifested urinary tract infection in our patient
urine leakage | first 3 days postoperative
  urine leakage from the percutaneous renal tract
irrigation fluid usage | intraoperative finding
  amount of irrigation fluid used during the surgery in liters
postoperative fever | first 2 days post surgery
  incidence of postoperative fever more than 38 c
need for DJ application | intraoperative finding
  the need for DJ application intraoperative due to rough manipulation, bleeding or residual stones
incidence of intraoperative colonic injury | intraoperative finding
  the accident injury to adjacent colon

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No